CLINICAL TRIAL: NCT03909997
Title: Severe Complications After Gastrectomy for Esophagogastric Junction and Gastric Cancer: Perioperative Results and Long Term Survival
Brief Title: Severe Complications After Gastrectomy for Esophagogastric Junction and Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Dr Sotero del Rio (Other)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2019-04-06; First posted 2019-04-10 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Gastric Cancer; Esophagogastric Junction Disorder
Keywords: Stomach neoplasms; gastrectomy; Risk factors; morbidity; adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gastrectomy is the main treatment for gastric and Siewert type II-III esophagogastric junction (EGJ) cancer. This surgery is associated with significant morbidity. The aim of the present study is to identify the predictors of postoperative morbidity and to evaluate long term survival according to complications. This is a retrospective cohort study.

DETAILED DESCRIPTION:
Gastrectomy is the main treatment for gastric and Siewert type II-III esophagogastric junction (EGJ) cancer. This surgery is associated with significant morbidity. The aim of the present study is to identify the predictors of postoperative morbidity and to evaluate long term survival according to complications.

This was a retrospective cohort study. The investigators included patients treated with gastrectomy for gastric or EGJ cancers at a single center. Severe morbidity was defined as Clavien-Dindo score ≥3.

The following factors are analyzed: age, sex, comorbidity, American Society of Anesthesiologists (ASA) physical status, tobacco and alcohol consumption, body mass index (BMI), hematocrit, serum albumin level, tumor location, the use of preoperative chemotherapy, laparoscopic or open surgery, total or subtotal gastrectomy, duodenal stump closure, multi-organ resection, lymphadenectomy, reconstruction method, T status, lymph node metastasis, and resection margin. The T stage was grouped by T1-T2 and T3-T4 for analysis. Patients will be followed for 5 years after surgery for survival analysis. A multivariate analysis is performed to identify predictors of overall and severe morbidity; and predictors of long-term survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with a gastrectomy for gastric cancer or esophagogastric cancer.
* Confirmed adenocarcinoma histology.

Exclusion Criteria:

* Histology different from adenocarcinoma.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive patients treated with a gastrectomy for gastric cancer or esophagogastric cancer at a single center are included.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-04-05 (Actual); Primary Completion 2021-04-05 (Estimated); Study Completion 2022-04-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients with severe 30-day or in-hospital morbidity | Perioperative
  Clavien 3 or higher complications

SECONDARY OUTCOMES:
Median and percentage of patients with long-term survival | 5 years
  5 year survival

CONTACTS AND LOCATIONS:
Overall Officials: Enrique M Norero, MD, Principal Investigator — Hospital Sotero Del Rio
Locations (1):
- Hospital Sotero del Rio, Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park DJ, Lee HJ, Kim HH, Yang HK, Lee KU, Choe KJ. Predictors of operative morbidity and mortality in gastric cancer surgery. Br J Surg. 2005 Sep;92(9):1099-102. doi: 10.1002/bjs.4952. PMID 15931657
- [Background] Onate-Ocana LF, Cortes-Cardenas SA, Aiello-Crocifoglio V, Mondragon-Sanchez R, Ruiz-Molina JM. Preoperative multivariate prediction of morbidity after gastrectomy for adenocarcinoma. Ann Surg Oncol. 2000 May;7(4):281-8. doi: 10.1007/s10434-000-0281-9. PMID 10819368
- [Background] Bartlett EK, Roses RE, Kelz RR, Drebin JA, Fraker DL, Karakousis GC. Morbidity and mortality after total gastrectomy for gastric malignancy using the American College of Surgeons National Surgical Quality Improvement Program database. Surgery. 2014 Aug;156(2):298-304. doi: 10.1016/j.surg.2014.03.022. Epub 2014 Mar 16. PMID 24947651
- [Background] Kim TH, Suh YS, Huh YJ, Son YG, Park JH, Yang JY, Kong SH, Ahn HS, Lee HJ, Slankamenac K, Clavien PA, Yang HK. The comprehensive complication index (CCI) is a more sensitive complication index than the conventional Clavien-Dindo classification in radical gastric cancer surgery. Gastric Cancer. 2018 Jan;21(1):171-181. doi: 10.1007/s10120-017-0728-3. Epub 2017 Jun 8. PMID 28597328
- [Background] Lee KG, Lee HJ, Yang JY, Oh SY, Bard S, Suh YS, Kong SH, Yang HK. Risk factors associated with complication following gastrectomy for gastric cancer: retrospective analysis of prospectively collected data based on the Clavien-Dindo system. J Gastrointest Surg. 2014 Jul;18(7):1269-77. doi: 10.1007/s11605-014-2525-1. Epub 2014 May 13. PMID 24820136
- [Background] Kikuchi H, Miyata H, Konno H, Kamiya K, Tomotaki A, Gotoh M, Wakabayashi G, Mori M. Development and external validation of preoperative risk models for operative morbidities after total gastrectomy using a Japanese web-based nationwide registry. Gastric Cancer. 2017 Nov;20(6):987-997. doi: 10.1007/s10120-017-0706-9. Epub 2017 Mar 11. PMID 28285387
- [Background] Norero E, Vega EA, Diaz C, Cavada G, Ceroni M, Martinez C, Briceno E, Araos F, Gonzalez P, Baez S, Vinuela E, Caracci M, Diaz A. Improvement in postoperative mortality in elective gastrectomy for gastric cancer: Analysis of predictive factors in 1066 patients from a single centre. Eur J Surg Oncol. 2017 Jul;43(7):1330-1336. doi: 10.1016/j.ejso.2017.01.004. Epub 2017 Feb 10. PMID 28359594
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Hayashi T, Yoshikawa T, Aoyama T, Ogata T, Cho H, Tsuburaya A. Severity of complications after gastrectomy in elderly patients with gastric cancer. World J Surg. 2012 Sep;36(9):2139-45. doi: 10.1007/s00268-012-1653-6. PMID 22610266
- [Background] Kim W, Kim HH, Han SU, Kim MC, Hyung WJ, Ryu SW, Cho GS, Kim CY, Yang HK, Park DJ, Song KY, Lee SI, Ryu SY, Lee JH, Lee HJ; Korean Laparo-endoscopic Gastrointestinal Surgery Study (KLASS) Group. Decreased Morbidity of Laparoscopic Distal Gastrectomy Compared With Open Distal Gastrectomy for Stage I Gastric Cancer: Short-term Outcomes From a Multicenter Randomized Controlled Trial (KLASS-01). Ann Surg. 2016 Jan;263(1):28-35. doi: 10.1097/SLA.0000000000001346. PMID 26352529
- [Background] Climent M, Hidalgo N, Vidal O, Puig S, Iglesias M, Cuatrecasas M, Ramon JM, Garcia-Albeniz X, Grande L, Pera M. Postoperative complications do not impact on recurrence and survival after curative resection of gastric cancer. Eur J Surg Oncol. 2016 Jan;42(1):132-9. doi: 10.1016/j.ejso.2015.08.163. Epub 2015 Sep 3. PMID 26385054
- [Background] Tokunaga M, Tanizawa Y, Bando E, Kawamura T, Terashima M. Poor survival rate in patients with postoperative intra-abdominal infectious complications following curative gastrectomy for gastric cancer. Ann Surg Oncol. 2013 May;20(5):1575-83. doi: 10.1245/s10434-012-2720-9. Epub 2012 Oct 18. PMID 23076557
- [Background] Kubota T, Hiki N, Sano T, Nomura S, Nunobe S, Kumagai K, Aikou S, Watanabe R, Kosuga T, Yamaguchi T. Prognostic significance of complications after curative surgery for gastric cancer. Ann Surg Oncol. 2014 Mar;21(3):891-8. doi: 10.1245/s10434-013-3384-9. Epub 2013 Nov 20. PMID 24254205

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT03909997/Prot_SAP_000.pdf